CLINICAL TRIAL: NCT07163988
Title: High-Sensitivity Cardiac Troponin I as a Diagnostic Marker for AMI Clinical Stage Classification in Acute Myocardial Infarction: A Retrospective Multicenter Study
Brief Title: Acute MI Staging Diagnosis by High-sensitivity Cardiac Troponin-I
Acronym: MIRON-4T
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other); Synergy Cardiovascular Research Center (Unknown)
Responsible Party: Principal Investigator, Keyur Vora, Director, Clinical Imaging Research Trials, Medical Imaging Research Institute, Indiana University School of Medicine
Other Study IDs: 27356b
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Hemorrhagic Myocardial Infarction; CCS-AMI Stages of Myocardial Infarction; High sensitivity Cardiac Troponin-I; Non-hemorrhagic Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Index STEMI with Primary PCI with Stenting: The study population consists of individuals aged 18 to 80 who have been diagnosed with acute ST-elevation myocardial infarction (STEMI) and are scheduled for emergency percutaneous coronary intervention (PCI).

SUMMARY:
MIRON-4T is a multicenter retrospective diagnostic study designed to evaluate the role of high-sensitivity cardiac troponin I (hs-cTnI) in the diagnosis and clinical stage classification of acute myocardial infarction as defined by the CCS-AMI staging system.

The study retrospectively analyzes biomarker data from patients diagnosed with AMI across multiple institutions, focusing on whether hs-cTnI levels-measured at specific time points-can reliably identify and stratify patients into CCS-defined AMI clinical stages (Stage 1 to Stage 4). It aims to correlate hs-cTnI kinetics and peak levels with clinical stage, presentation patterns, and outcomes.

This trial seeks to offer a biomarker-based alternative to imaging-heavy staging, potentially streamlining early diagnosis and therapeutic triage for AMI patients in varied clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 years
* Index STEMI
* Coronary angiogram with PCI to occur irrespective of the onset of the symptoms.
* Ability to provide informed consent for themselves

Exclusion Criteria:

* History of prior myocardial infarction,
* Cardiogenic shock,
* Patients who present with current cardiac arrest
* Any contraindication to cardiac CMR (claustrophobia, pacemaker or cardiac defibrillator, known allergy to gadolinium),
* Presence of permanent atrial fibrillation,
* Unconscious patient,
* Severe renal insufficiency (creatinine clearance ≤ 30 ml/min/m2 or renal replacement therapy),
* Women who are pregnant or breastfeeding. Women of reproductive potential must have a negative pregnancy test.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged 18 to 80 who have been diagnosed with acute ST-elevation myocardial infarction (STEMI) and are scheduled for emergency percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
High-sensitivity Cardiac Troponin-I Thresholds | 48 hours
  Levels of hs-cTn-I to differentiate AMI Stages I-IV (Classified by CMR)
Time window for high-sensitivity cardiac troponin-I thresholds | 48 hours
  Define time window for high-sensitivity cardiac troponin-I threshold for AMI Stages I-IV

SECONDARY OUTCOMES:
Adjusted Risk Ratio | 48 hours
  Adjusted Risk Ratio to explore parameters to predict AMI Stages I-IV

CONTACTS AND LOCATIONS:
Locations (2):
- Medical Imaging Research Institute, Indianapolis, Indiana, United States
- Synergy Cardiovascular Research Center, Rajkot, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vora KP, Kalra A, Shah CD, Bhatt K, Kumar A, Pandya T, Poptani V, Chan SF, Singh D, Jambunathan N, Subramanian R, Youssef K, Kanakasabai S, Finney R, Desai A, Kreutz RP, Kovacs RJ, Raman SV, Bhatt DL, Dharmakumar R. In-Hospital Mortality in Hemorrhagic Myocardial Infarction. NEJM Evid. 2025 Sep;4(9):EVIDoa2400294. doi: 10.1056/EVIDoa2400294. Epub 2025 Aug 26. PMID 40858097
- [Background] Vora KP, Kumar A, Krishnam MS, Prato FS, Raman SV, Dharmakumar R. Microvascular Obstruction and Intramyocardial Hemorrhage in Reperfused Myocardial Infarctions: Pathophysiology and Clinical Insights From Imaging. JACC Cardiovasc Imaging. 2024 Jul;17(7):795-810. doi: 10.1016/j.jcmg.2024.02.003. Epub 2024 Apr 10. PMID 38613553
- [Background] Kumar A, Connelly K, Vora K, Bainey KR, Howarth A, Leipsic J, Betteridge-LeBlanc S, Prato FS, Leong-Poi H, Main A, Atoui R, Saw J, Larose E, Graham MM, Ruel M, Dharmakumar R. The Canadian Cardiovascular Society Classification of Acute Atherothrombotic Myocardial Infarction Based on Stages of Tissue Injury Severity: An Expert Consensus Statement. Can J Cardiol. 2024 Jan;40(1):1-14. doi: 10.1016/j.cjca.2023.09.020. Epub 2023 Oct 28. PMID 37906238